CLINICAL TRIAL: NCT02034994
Title: Combining Primary and Secondary Prevention for Reduction of Excessive Weight Gain in School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, MD, PhD. Full Professor of Epidemiology, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMS-PAPPAS2-project
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: school-based intervention; after school physical activity; sugar sweetened beverages; sedentary behavior; schoolchildren
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Reduction of sugar sweetened beverages. cookies, sedentary activities and increasing physical activity
  Interventions: Behavioral: Eating behavior and physical activity change
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Eating behavior and physical activity change — A combination of two prevention school based programs will be addressed to schoolchildren over one year. Primary prevention will be developed monthly in order to reduce cookies and sugar sweetened beverages consumption, reduction of sedentary activities, increase meal consumption frequency and quality etc, in all children from 6th and 7th grades. Overweight and obese children will be invited to participate on a secondary prevention program in which daily physical activity classes will be performed by physical education teachers in school facilities.
  Arms: Intervention group

SUMMARY:
The main objective is to evaluate the effects of a multicomponent, school-based intervention combining change in nutritional behaviors with after school physical activity activities in reducing the excessive weight gain in schoolchildren.

DETAILED DESCRIPTION:
Specific objectives are:

- evaluate the effect of the program on: change in nutritional behaviors, such as reducing sugar sweetened beverages and cookies intake reduction of time spent in sedentary activities gains in school performance and cognition outcomes the amount of daily physical activity on the percentage of body fat, changes in biochemical markers and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

Both prevention programs:

* 6th and 7th grades students
* consent form signed by parents / tutors

Secondary prevention program:

- overweight and obese children

Exclusion Criteria:

* pregnant girls

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2014-02-15 (Actual); Primary Completion 2014-11-15 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | One Year

SECONDARY OUTCOMES:
Mean lean and fatty body mass proportions: measured by portable electrical bioimpedance bean | One year

OTHER OUTCOMES:
Sedentary activities | One year
Sugar sweetened beverages intake | one year
cookies intake | one year
fruits intake | one year
physical activity | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Public Schools, Niterói, Rio de Janeiro, Brazil